CLINICAL TRIAL: NCT00085202
Title: Treatment of Patients With Newly Diagnosed Medulloblastoma, Supratentorial Primitive Neuroectodermal Tumor, or Atypical Teratoid Rhabdoid Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJMB03; NCI-2011-01185 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma; untreated childhood supratentorial primitive neuroectodermal tumor; childhood atypical teratoid/rhabdoid tumor; untreated childhood pineoblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Rhabdoid Tumor | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum 1 (high-risk group) (Experimental): Patients undergo craniospinal radiotherapy once daily 5 days a week for 6 weeks. Six weeks after the completion of radiotherapy, patients receive high-dose chemotherapy followed by autologous stem cell transplantation (SCT) and filgrastim (G-CSF) with post-transplantation vincristine. High-dose chemotherapy and autologous SCT repeat every 4 weeks for 3 additional courses in the absence of unacceptable toxicity.
  Interventions: vincristine, cisplatin, cyclophosphamide, autologous hematopoietic stem cell transplantation, filgrastim, radiation therapy
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: vincristine; Procedure: autologous hematopoietic stem cell transplantation; Radiation: radiation therapy
- Stratum 2 (average-risk group) (Experimental): Patients undergo craniospinal radiotherapy as in stratum 1, but at a lower dose. Patients receive high-dose chemotherapy, autologous SCT, G-CSF, and post-transplantation vincristine as in stratum 1.
  Interventions: vincristine, cisplatin, cyclophosphamide, autologous hematopoietic stem cell transplantation, filgrastim, radiation therapy
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: vincristine; Procedure: autologous hematopoietic stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given subcutaneously
  Other Names: Neupogen(R); G-CSF
Drug: cisplatin — Given IV
  Other Names: Platinol-AQ(R)
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan(R)
Drug: vincristine — Given IV
  Other Names: Oncovin(R)
Procedure: autologous hematopoietic stem cell transplantation — Patients undergo autologous stem cell transplantation
  Other Names: autologous HSCT
Radiation: radiation therapy — Patients undergo craniospinal radiotherapy once daily 5 days a week for 6 weeks.
  Other Names: RT; Craniospinal radiotherapy

SUMMARY:
Drugs used in chemotherapy, such as vincristine, cisplatin, and cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. Autologous stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy or radiation therapy. It is not yet known which radiation therapy regimen combined with chemotherapy and donor stem cell transplant is more effective in treating medulloblastoma, supratentorial primitive neuroectodermal tumor, or atypical teratoid rhabdoid tumor.

This phase III trial is studying two different regimens of radiation therapy when given together with chemotherapy and autologous stem cell transplant to see how well they work in treating patients with newly diagnosed medulloblastoma, supratentorial primitive neuroectodermal tumor, or atypical teratoid rhabdoid tumor.

PRIMARY OBJECTIVE:

* To assess the relationship between ERBB2 protein expression in tumors and progression-free survival probability for patients with medulloblastoma.
* To estimate the frequency of mutations associated with SHH and WNT tumors (as defined by gene expression profiling) via targeted sequencing performed in an independent cohort of WNT and SHH tumors (also defined by gene expression profiling).

DETAILED DESCRIPTION:
SECONDARY OBJECTIVES:

* To compare the effects of a computer-based training system specifically targeting language, reading, and learning skills (Fast ForWord, Scientific Learning Corporation) with the current standard of care on reading decoding skills as measured by individual academic testing.
* To monitor for treatment failure in the posterior fossa of patients whose tumor bed receives a reduced volume of radiation.
* To correlate radiation dosimetry of target and normal tissues with rate and patterns of failure and longitudinal measures of audiometric, endocrine and cognitive effects.

EXPLORATORY OBJECTIVES:

* To estimate the change in neuropsychological performance from the neuropsychology assessment battery (intellect, academic achievement and cognitive ability) and examine the relationship of these changes to risk group, age at diagnosis, and parent measures.
* To evaluate the differences between neurotoxicity in the average-risk patient group with that in the high-risk group through qMRI, and fMRI.
* To develop or refine novel models relating impact of medulloblastoma therapy on neurocognitive performance to quantitative and functional neuroimaging measures.

OUTLINE: This is a multicenter study. Patients are stratified according to disease risk (high-risk disease vs average-risk disease).

Patients in both strata undergo peripheral blood stem cell or bone marrow harvest.

* Stratum 1 (high-risk group):

  * Radiotherapy: Patients undergo craniospinal radiotherapy once daily 5 days a week for 6 weeks.
  * High-dose chemotherapy and autologous stem cell transplantation (SCT): Six weeks after the completion of radiotherapy, patients receive high-dose chemotherapy comprising vincristine IV followed by cisplatin IV over 6 hours on day -4 and cyclophosphamide IV over 1 hour on days -3 and -2. Patients undergo autologous SCT on day 0. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 1 and continuing until blood counts recover. Patients receive vincristine IV on day 6. High-dose chemotherapy and autologous SCT repeat every 4 weeks for 3 additional courses in the absence of unacceptable toxicity.
* Stratum 2 (average-risk group):

  * Radiotherapy: Patients undergo craniospinal radiotherapy as in stratum 1, but at a lower dose.
  * High-dose chemotherapy and autologous SCT: Patients receive high-dose chemotherapy, autologous SCT, G-CSF, and post-transplantation vincristine as in stratum 1.

Some patients undergo a neuropsychology assessment at baseline, before chemotherapy, and then annually for 5 years.

After completion of study therapy, patients are followed every 3 months until month 30 (2.5 years) after diagnosis and then every 6 months until month 72 (6 years) after diagnosis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Medulloblastoma
  * Supratentorial primitive neuroectodermal tumor (PNET)
  * PNET variants (ependymoblastoma, pineoblastoma, CNS neuroblastoma)
  * Atypical teratoid rhabdoid tumor (ATRT)
* Definitive surgery for CNS tumor within the past 31 days
* Meets one of the following risk criteria:

  * Average-risk disease

    * Localized disease with no overt evidence of invasion beyond the posterior fossa (or supratentorial compartment for PNET or ATRT) by intraoperative observations of the neurosurgeon AND postoperative CT scan or MRI
    * T4 disease eligible if all of the following are true:

      * Gross total resection determined by intraoperative observations of the neurosurgeon AND postoperative CT scan or MRI
      * Residual tumor or imaging abnormality whose size is < 1.5 cm^2
      * No evidence of CNS or extraneural metastasis by MRI of the spine (with and without contrast agent) or CT-based myelogram AND by cytologic examination of the lumbar cerebral spinal fluid (CSF) 14-28 days after surgery
    * Brain stem invasion allowed in the absence of residual tumor (tumor < 1.5 cm^2 by imaging)
  * High-risk disease meeting one of the following criteria:

    * Metastatic disease within the neuraxis (i.e., evidence of subarachnoid dissemination by imaging and/or cytologic examination of CSF)
    * Presence of residual disease > 1.5 cm^2 at the primary site after surgery

PATIENT CHARACTERISTICS:

Age

* 3 to 21 at diagnosis

Performance status

* Lansky 30-100% (< 10 years old)
* Karnofsky 30-100% (≥ 10 years old) (except for posterior fossa syndrome)

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 8 g/dL
* WBC > 2,000/mm^3
* Absolute neutrophil count > 500/mm^3
* Platelet count > 50,000/mm^3

Hepatic

* ALT < 5 times normal
* Bilirubin < 3.0 mg/dL

Renal

* Creatinine < 2.0 mg/dL OR
* Creatinine clearance > 70 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Prior corticosteroid therapy allowed

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 416 (Actual)
Dates: Start 2003-08; Primary Completion 2016-12 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (9):
- United States (4):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Lady Cilento Children's Hospital, Brisbane, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Acharya S, Guo Y, Patni T, Li Y, Wang C, Gargone M, Ashford JM, Wilson L, Faught A, Reddick WE, Patay Z, Gajjar A, Conklin HM, Merchant TE. Association Between Brain Substructure Dose and Cognitive Outcomes in Children With Medulloblastoma Treated on SJMB03: A Step Toward Substructure-Informed Planning. J Clin Oncol. 2022 Jan 1;40(1):83-95. doi: 10.1200/JCO.21.01480. Epub 2021 Oct 29. PMID 34714708
- [Derived] Partanen M, Anghelescu DL, Hall L, Schreiber JE, Rossi M, Gajjar A, Jacola LM. Longitudinal associations between exposure to anesthesia and neurocognitive functioning in pediatric medulloblastoma. Eur J Cancer. 2021 May;148:103-111. doi: 10.1016/j.ejca.2021.02.010. Epub 2021 Mar 17. PMID 33743477
- [Derived] Kumar R, Smith KS, Deng M, Terhune C, Robinson GW, Orr BA, Liu APY, Lin T, Billups CA, Chintagumpala M, Bowers DC, Hassall TE, Hansford JR, Khuong-Quang DA, Crawford JR, Bendel AE, Gururangan S, Schroeder K, Bouffet E, Bartels U, Fisher MJ, Cohn R, Partap S, Kellie SJ, McCowage G, Paulino AC, Rutkowski S, Fleischhack G, Dhall G, Klesse LJ, Leary S, Nazarian J, Kool M, Wesseling P, Ryzhova M, Zheludkova O, Golanov AV, McLendon RE, Packer RJ, Dunham C, Hukin J, Fouladi M, Faria CC, Pimentel J, Walter AW, Jabado N, Cho YJ, Perreault S, Croul SE, Zapotocky M, Hawkins C, Tabori U, Taylor MD, Pfister SM, Klimo P Jr, Boop FA, Ellison DW, Merchant TE, Onar-Thomas A, Korshunov A, Jones DTW, Gajjar A, Ramaswamy V, Northcott PA. Clinical Outcomes and Patient-Matched Molecular Composition of Relapsed Medulloblastoma. J Clin Oncol. 2021 Mar 1;39(7):807-821. doi: 10.1200/JCO.20.01359. Epub 2021 Jan 27. PMID 33502920
- [Derived] Gajjar A, Robinson GW, Smith KS, Lin T, Merchant TE, Chintagumpala M, Mahajan A, Su J, Bouffet E, Bartels U, Schechter T, Hassall T, Robertson T, Nicholls W, Gururangan S, Schroeder K, Sullivan M, Wheeler G, Hansford JR, Kellie SJ, McCowage G, Cohn R, Fisher MJ, Krasin MJ, Stewart CF, Broniscer A, Buchhalter I, Tatevossian RG, Orr BA, Neale G, Klimo P Jr, Boop F, Srinivasan A, Pfister SM, Gilbertson RJ, Onar-Thomas A, Ellison DW, Northcott PA. Outcomes by Clinical and Molecular Features in Children With Medulloblastoma Treated With Risk-Adapted Therapy: Results of an International Phase III Trial (SJMB03). J Clin Oncol. 2021 Mar 1;39(7):822-835. doi: 10.1200/JCO.20.01372. Epub 2021 Jan 6. PMID 33405951
- [Derived] Xu H, Robinson GW, Huang J, Lim JY, Zhang H, Bass JK, Broniscer A, Chintagumpala M, Bartels U, Gururangan S, Hassall T, Fisher M, Cohn R, Yamashita T, Teitz T, Zuo J, Onar-Thomas A, Gajjar A, Stewart CF, Yang JJ. Common variants in ACYP2 influence susceptibility to cisplatin-induced hearing loss. Nat Genet. 2015 Mar;47(3):263-6. doi: 10.1038/ng.3217. Epub 2015 Feb 9. PMID 25665007
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 416 participants were enrolled between 9/9/2003 and 3/7/2013.
Pre-assignment Details: Of the 416 participants enrolled, three were ineligible and taken off study.
Groups:
- Average-Risk Group: Participants assigned to the average-risk arm had localized tumor without overt evidence of invasion beyond the posterior fossa (or supratentorial compartment for PNET's/ATRT). Participants with T4 disease met the following criteria: gross total resection defined as residual tumor or imaging abnormality whose size was <1.5 cm^2 on postoperative CT or MR images, no evidence of CNS or extraneural metastasis, and brain stem invasion by the tumor in the absence of imaging evidence of residual tumor (tumor size <1.5 cm^2).
- High-Risk Group: Participants assigned to the high-risk arm were determined to have the presence of metastatic disease within the neuraxis (i.e., evidence of subarachnoid dissemination), OR presence of residual disease (≥1.5 cm^2) at the primary site after surgery.
Period: Overall Study
Arm/Group | Average-Risk Group | High-Risk Group
Started | 269 | 144
Completed | 251 | 120
Not Completed | 18 | 24
Not completed — Still on therapy | 2 | 0
Not completed — Bone involvement confirmed by bone scan | 0 | 1
Not completed — Excessive toxicity | 6 | 5
Not completed — Non-specified | 3 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Progressive disease | 1 | 11

BASELINE CHARACTERISTICS:
Population: Participants had a diagnosis of medulloblastoma, supratentorial primitive neuroectodermal tumor (PNET), PNET variants (ependymoblastoma, pineoblastoma, CNS neuroblastoma), or atypical teratoid rhabdoid tumor (ATRT).
Groups:
- Total: Total of all reporting groups
Arm/Group | Average-Risk Group | High-Risk Group | Total
Number analyzed (Participants) | 269 | 144 | 413
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.15 (4.08) | 8.66 (3.93) | 8.98 (4.03)
Age, Continuous [Median (Full Range); unit: years] | 8.42 [3.06 to 21.56] | 7.87 [3.13 to 20.43] | 8.33 [3.06 to 21.56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 56 | 161
  Male | 164 | 88 | 252

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in ERBB2-Negative Tumors Compared to ERBB2-Positive Tumors
Description: The relationship between ERBB2 protein expression in tumors and progression-free survival was assessed in 122 participants with a diagnosis of medulloblastoma and with ERBB2 protein assessments. If the ERBB2 value was greater than zero, the ERBB2 was defined as positive for the participant. If the ERBB2 value was zero, the ERBB2 was defined as negative. Progression-free survival was calculated from the date of diagnosis to the date of disease progression/relapse, the date of death, or the date of last contact. The log-rank test was used to compare the PFS distributions of ERBB2 groups.
Time Frame: 2 years after tumor cell analysis in 122 participants
Population: Analysis included the first 122 participants with a diagnosis of medulloblastoma and with fresh tissue and ERBB2 protein assessments. Participants with a diagnosis of PNET, PNET variants, or ATRT were not included in this analysis.
Measure: Number (95% Confidence Interval); unit: probability of PFS at 2 years
Groups:
- Overall Study: Analysis included the first 122 participants with a diagnosis of medulloblastoma and with fresh tissue and ERBB2 protein assessments. Participants with a diagnosis of supratentorial primitive neuroectodermal tumor (PNET), PNET variants (ependymoblastoma, pineoblastoma, CNS neuroblastoma), or atypical teratoid rhabdoid tumor (ATRT) were not included in the analysis of ERBB2 tumors.
- Average-Risk Group: Participants assigned to the average-risk arm had localized tumor without overt evidence of invasion beyond the posterior fossa. Participants with T4 disease met the following criteria: gross total resection defined as residual tumor or imaging abnormality whose size was <1.5 cm^2 on postoperative CT or MR images, no evidence of CNS or extraneural metastasis, and brain stem invasion by the tumor in the absence of imaging evidence of residual tumor (tumor size <1.5 cm^2).
Arm/Group | Overall Study | Average-Risk Group | High-Risk Group
Number analyzed (Participants) | 122 | 85 | 37
probability of PFS at 2 years
  Positive ERBB2: number analyzed (Participants) | 77 | 54 | 23
  Positive ERBB2 | 79.2 [70.4 to 88.0] | 83.3 [73.5 to 93.1] | 69.6 [50.8 to 88.4]
  Negative ERBB2: number analyzed (Participants) | 45 | 31 | 14
  Negative ERBB2 | 86.7 [76.9 to 96.5] | 93.5 [85.1 to 100] | 71.4 [48.9 to 93.9]
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p = 0.8001, Log Rank
Statistical Analysis 2: Comparison: Average-Risk Group; Test type: Superiority or Other; p = 0.5195, Log Rank
Statistical Analysis 3: Comparison: High-Risk Group; Test type: Superiority or Other; p = 0.7696, Log Rank

2. Primary Outcome: Progression-Free Survival (PFS) Compared Between ERBB2 Assessment and Risk Group.
Description: 122 participants with a diagnosis of medulloblastoma were grouped by ERBB2 positive/negative assessment and risk group into 4 groups. Progression-free survival was calculated from the date of diagnosis to the date of disease progression/relapse, the date of death, or the date of last contact. The log-rank test was used to compare the PFS distributions of ERBB2 groups.
Time Frame: 2 years after tumor cell analysis in 122 participants
Population: Analysis was completed for the first 122 participants with a diagnosis of medulloblastoma and with fresh tissue and ERBB2 protein assessments. Participants with a diagnosis of PNET, PNET variants, or ATRT were not included in this analysis.
Measure: Number (95% Confidence Interval); unit: probability of PFS at 2 years
Groups:
- ERBB2 Positive & Average Risk: 54 participants who were ERBB2 positive and in the average risk group.
- ERBB2 Positive & High Risk: 23 participants who were ERBB2 positive and in the high risk group
- ERBB2 Negative & Average Risk: 31 participants who were ERBB2 negative and in the average risk group
- ERBB2 Negative & High Risk: 14 participants who were ERBB2 negative and in the high risk group
Arm/Group | ERBB2 Positive & Average Risk | ERBB2 Positive & High Risk | ERBB2 Negative & Average Risk | ERBB2 Negative & High Risk
Number analyzed (Participants) | 54 | 23 | 31 | 14
probability of PFS at 2 years | 83.3 [73.5 to 93.1] | 69.6 [50.8 to 88.4] | 93.5 [85.1 to 100] | 71.4 [48.9 to 93.9]
Statistical Analysis 1: Comparison: ERBB2 Positive & Average Risk vs ERBB2 Positive & High Risk vs ERBB2 Negative & Average Risk vs ERBB2 Negative & High Risk; Test type: Superiority or Other; p = 0.0206, Log Rank

3. Primary Outcome: Frequency of Mutations Associated With SHH and WNT Tumors
Description: The frequency of mutations for the main genes associated with SHH and WNT tumors identified via targeted sequencing based on formalin fixed paraffin embedded material is provided.
Time Frame: within 3.5 years following completion of accrual
Population: Only patients with WNT and SHH tumors with available tissue for targeted sequencing were analyzed for frequency of mutation. WNT and SHH subgroups were identified by methylation profiling.
Measure: Count of Participants; unit: Participants
Groups:
- SHH Pathway - In/Del Somatic; WNT Pathway - In/Del Somatic: Tissue from this subgroup of patients was analyzed for somatic insertion/deletion (In/Del).
- SHH Pathway - In/Del Germline; WNT Pathway - In/Del Germline: Tissue from this subgroup of patients was analyzed for germline insertion/deletion (In/Del).
- SHH Pathway - SNV Somatic; WNT Pathway - SNV Somatic: Tissue from this subgroup of patients was analyzed for somatic single nucleotide variation (SNV).
- SHH Pathway - SNV Germline; WNT Pathway - SNV Germline: Tissue from this subgroup of patients was analyzed for germline single nucleotide variation (SNV).
Arm/Group | SHH Pathway - In/Del Somatic | WNT Pathway - In/Del Somatic | SHH Pathway - In/Del Germline | WNT Pathway - In/Del Germline | SHH Pathway - SNV Somatic | WNT Pathway - SNV Somatic | SHH Pathway - SNV Germline | WNT Pathway - SNV Germline
Number analyzed (Participants) | 20 | 18 | 20 | 18 | 20 | 18 | 20 | 18
Participants
  PTCH1 | 7 | 0 | 0 | 0 | 4 | 0 | 0 | 0
  DDX3X | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 0
  TP53 | 0 | 0 | 0 | 0 | 5 | 3 | 0 | 0
  KMT2D | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  SUFU | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREBBP | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  GLI2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  TCF4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PTEN | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
  KMT2C | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
  FBXW7 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
  GSE1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CTNNB1 | 0 | 0 | 0 | 0 | 1 | 18 | 0 | 0
  SMARCA4 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
  PIK3CA | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  APC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  EPHA7 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ARID1A | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  ARID2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ATM | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BRCA2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Reading Decoding Composite Scores in the Intervention and Standard of Care Groups
Description: SOC is standard-of-Care control group. Patients randomly assigned to the control group received the current standard of care. RI is Reading Intervention Group. Patients randomly assigned to Reading Intervention Group which is with The Fast ForWord program. Assessment of reading decoding was completed using the Woodcock Johnson, Third Edition (WJIII) Tests of Achievement (Woodcock, McGraw, & Mather, 2001), with particular attention given to the reading and reading-related abilities. Two subtests were completed: (1) Letter-Word Identification, and (2) Word Attack, a test requiring the patient to read phonologically regular nonwords. The combination of these two subtests provided a standardized composite score of overall reading decoding ability with a population mean of 100 and a standard deviation of 15. Scores of 90-110 are considered to be in the average range, while those 80-89 are considered low-average (refer: Journal of Pediatric Psychology 39(4) pp. 450-458, 2014).
Time Frame: 5 years postdiagnosis
Population: Of the 126 MB patients enrolled, 41 were not eligible. This left 85 patients considered eligible for the randomization study. Of the 85 eligible patients,81 were randomized to either SOC (n= 38) or to RI (n =43). The parents of only four patients did not consent to the intervention study. Two patients randomized to the RI group, and four patients in the SOC group, were excluded due to having only a single assessment, which resulted in 75 patients (RI=41, SOC=34) over a 5-year follow-up period.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Intervention: A COMPUTER-BASED TRAINING SYSTEM SPECIFICALLY TARGETING LANGUAGE, READING, AND LEARNING SKILLS (FAST FORWORD®, SCIENTIFIC LEARNING CORPORATION)
- Standard of Care: THE CURRENT STANDARD OF CARE ON READING DECODING SKILLS
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 41 | 34
score on a scale
  Baseline | 104.1 (1.902) | 102.4 (2.604)
  Change over time | -1.51 (0.4849) | -1.17 (0.4883)
Statistical Analysis 1: Comparison: Intervention vs Standard of Care; Change over time; Test type: Superiority; p = 0.6231, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention vs Standard of Care; Baseline; Test type: Superiority; p = 0.5720, t-test, 2 sided

5. Secondary Outcome: Number of Average Risk Patients Whose Treatment Failure Included the Posterior Fossa
Description: To monitor for treatment failure in the posterior fossa of patients whose tumor bed receives a reduced volume of radiation.
Time Frame: Annually for 6 years post irradiation
Population: Analysis included 100 average risk participants with a diagnosis of medulloblastoma who had cumulative radiotherapy dose profiles and treatment failure volumes data available. All participants included in analysis who were still at risk and on-study were followed for a minimum of 6 years. Participants with a diagnosis of PNET, PNET variants, or ATRT were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Average-Risk Group
Number analyzed (Participants) | 100
Participants | 6

6. Secondary Outcome: Associative Memory for Two Risk Group at Enrollment
Description: Assessment of associative memory at enrollment. Associate memory score is a representative measurement of learning and recalling pictograph representations of words. It measures associative memory (Long-Term Retrieval). Mean=100, SD=15, Average Range 85-115. Higher is better.
Time Frame: At enrollment
Population: Children with medulloblastoma who were age 3-21 years at diagnosis and were enrolled on SJMB03 at St Jude Children's Research Hospital. Patients were excluded if the cumulative RT plan (Craniospinal Irradiation (CSI) and boost) could not be retrieved; if the baseline preRT Magnetic Resonance Image (MRI) scan was of poor quality, preventing delineation of brain substructures ; or if the patient had completed fewer than two specific neurocognitive evaluations for this objective.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Average Risk Group: Average-Risk Participants assigned to the average-risk arm had localized tumor without overt evidence of invasion beyond the posterior fossa. Participants with T4 disease met the following criteria: gross total resection defined as residual tumor or imaging abnormality whose size was <1.5 cm^2 on postoperative CT or MR images, no evidence of CNS or extraneural metastasis, and brain stem invasion by the tumor in the absence of imaging evidence of residual tumor (tumor size <1.5 cm^2).
- High Risk Group: Participants assigned to the high- risk arm were determined to have the presence of metastatic disease within the neuraxis (i.e., evidence of subarachnoid dissemination), OR presence of residual disease (≥1.5 cm^2) at the primary site after surgery.
Arm/Group | Average Risk Group | High Risk Group
Number analyzed (Participants) | 51 | 23
score on a scale | 93.61 (22.25) | 98.04 (18.56)

7. Secondary Outcome: Associative Memory for Two Risk Group at 5 Years After Enrollment
Description: Assessment of associative memory at 5 years after enrollment. Assessment of associative memory score at enrollment. Associate memory score is a representative measurement of learning and recalling pictograph representations of words. It measures associative memory (Long-Term Retrieval). Mean=100, SD=15, Average Range 85-115. Higher is better.
Time Frame: At 5 years after enrollment
Population: Children with medulloblastoma who were age 3-21 years at diagnosis and were enrolled on SJMB03 at St Jude Children's Research Hospital. Patients were excluded if the cumulative RT plan (Craniospinal Irradiation (CSI) and boost) could not be retrieved; if the baseline preRT Magnetic Resonance Image (MRI) scan was of poor quality, preventing delineation of brain substructures; or if the patient had completed fewer than two specific neurocognitive evaluations for this objective.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Average Risk Group | High Risk Group
Number analyzed (Participants) | 59 | 24
score on a scale | 98.73 (16.94) | 93.58 (13.7)

8. Secondary Outcome: Processing Speed for Two Risk Group at Enrollment
Description: Assessment of Processing Speed at enrollment. This score measure of Processing Speed based on Visual Matching and Decision Speed tests. Mean=100, SD=15, Average Range 85-115. Higher is better.
Time Frame: At enrollment
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Average Risk Group | High Risk Group
Number analyzed (Participants) | 48 | 21
score on a scale | 83.98 (18.53) | 87.29 (19.73)

9. Secondary Outcome: Processing Speed for Two Risk Group at 5 Years After Enrollment
Description: Assessment of Processing Speed at 5 years after enrollment. This score measure of Processing Speed based on Visual Matching and Decision Speed tests. Mean=100, SD=15, Average Range 85-115. Higher is better.
Time Frame: At 5 years after enrollment
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Average Risk Group | High Risk Group
Number analyzed (Participants) | 57 | 24
score on a scale | 84.21 (24.36) | 75.71 (25.71)

10. Secondary Outcome: Perceptual Speed for Two Risk Group at Enrollment
Description: Assessment of Perceptual Speed at enrollment. It measures rapidly locating and circling identical numbers from a set of numbers which reflects perceptual speed. Mean=100, SD=15, Average Range 85-115. Higher is better.
Time Frame: At enrollment
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Average Risk Group | High Risk Group
Number analyzed (Participants) | 49 | 23
score on a scale | 82.06 (19.99) | 90.04 (18.23)

11. Secondary Outcome: Perceptual Speed for Two Risk Group at 5 Years After Enrollment
Description: Assessment of Perceptual Speed at 5 years after enrollment. It measures rapidly locating and circling identical numbers from a set of numbers which reflects perceptual speed. Mean=100, SD=15, Average Range 85-115. Higher is better.
Time Frame: At 5 years after enrollment
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Average Risk Group | High Risk Group
Number analyzed (Participants) | 59 | 24
score on a scale | 78.68 (21.58) | 72.29 (27.32)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported through 9/17/2013 and include all grade 3, 4 and 5 events occurring during treatment to 30 days after treatment end, and events occurring >30 days after treatment end and felt to be possibly related to protocol treatment.
Description: Per protocol, Grade 3 and 4 hematologic toxicities, grade 3 and 4 electrolyte abnormalities, and total parenteral nutrition or intravenous fluids administered to prevent significant weight loss/malnutrition were not collected if they occurred from the beginning of radiation therapy through the end of 4 courses of high dose chemotherapy.
Arm/Group | Average-Risk Group | High-Risk Group
Serious Adverse Events (participants affected / at risk) | 17/269 | 17/144
Other Adverse Events (participants affected / at risk) | 236/269 | 118/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Average-Risk Group (N=269) | High-Risk Group (N=144)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia - sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac general - other (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Vascular disorders) | 0 (0) | 1 (1) — e.g., thrombotic thrombocytopenic purpura (TTP) or hemolytic uremic syndrome (HUS)
Death not associated with CTCAE term, death NOS (General disorders) | 0 (0) | 1 (1)
Hemorrhage/bleeding - other (Vascular disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 2 (2) | 0 (0) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L).
Infection, blood (Infections and infestations) | 1 (1) | 0 (0) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection with normal ANC or Grade 1 or 2 neutrophils, blood (Infections and infestations) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, meninges (meningitis) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, wound (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC, meninges (meningitis) (Infections and infestations) | 2 (2) | 0 (0)
Infection with unknown ANC, wound (Infections and infestations) | 0 (0) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Apnea (Nervous system disorders) | 0 (0) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 1 (1)
CNS necrosis/cystic progression (Nervous system disorders) | 1 (1) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 0 (0) | 2 (2)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Personality/behavioral (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 3 (3)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary/upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Syndromes - other (General disorders) | 1 (1) | 1 (1)
Pain - other (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Average-Risk Group (N=269) | High-Risk Group (N=144)
Febrile neutropenia (Infections and infestations) | 172 (383) | 77 (148) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L).
Infection, blood (Infections and infestations) | 55 (76) | 24 (28) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Vomiting (Gastrointestinal disorders) | 53 (63) | 21 (29)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 39 (54) | 23 (32)
Pain, abdomen NOS (General disorders) | 33 (37) | 17 (30)
Nausea (Gastrointestinal disorders) | 27 (30) | 20 (23)
Infection - other (Infections and infestations) | 25 (33) | 16 (19)
Diarrhea (Gastrointestinal disorders) | 23 (36) | 14 (16)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 22 (28) | 7 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils, blood (Infections and infestations) | 21 (30) | 9 (11)
Anorexia (Gastrointestinal disorders) | 17 (17) | 12 (13)
Infection with unknown ANC, blood (Infections and infestations) | 17 (23) | 13 (19)
Infection with normal ANC or Grade 1 or 2 neutrophils, catheter-related (Infections and infestations) | 16 (21) | 3 (3)
Hypotension (Cardiac disorders) | 16 (17) | 14 (19)
Hypertension (Cardiac disorders) | 15 (25) | 10 (12)
Infection, catheter-related (Infections and infestations) | 14 (15) | 5 (7) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Hemorrhage, pulmonary/upper respiratory, nose (Vascular disorders) | 14 (20) | 11 (16)
Pain, head/headache (General disorders) | 13 (13) | 10 (14)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 11 (12) | 9 (9)

LIMITATIONS AND CAVEATS:
The study participants for Secondary Outcome Measure #4 were randomized to standard-of-care group vs. reading intervention after medical treatment. The participants were a subset of patients who contributed to the primary aim and who signed a separate consent form distinct from the main medical treatment consent. They were then randomly assigned to either the standard-of-care group (SOC) or to the reading intervention (RI) group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes